CLINICAL TRIAL: NCT03204292
Title: Measurement of the Inferior Vena Cava as a Method of Evaluating the Fluid Balance of Mechanically Ventilated Patients
Brief Title: Evaluating the Fluid Balance of Mechanically Ventilated Patients by Ultrasonography
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, senior assistant, Jagiellonian University
Other Study IDs: 122.6120.85.2015
Record Dates: First submitted 2017-06-24; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Fluid Overload; Fluid Loss
Keywords: Inferior vena cava; Fluid responsiveness; Central venous pressure
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IVC/Ao: ultrasound, the inferior vena cava and abdominal aorta were measured. Inferior vena cava width was assessed at an interval of approximately 1 cm distal from connection of the hepatic vein to the inferior vena cava. No significant changes were observed in the width of the inferior vena cava during various respiratory phases, because of the positive pressure ventilation. The widest value was always chosen for the data. The assessment of the width of the abdominal aorta was performed above arise of the celiac trunk, at the height of the vein of the lower vena cava.

SUMMARY:
ratio of the diameter of inferior vena cava to the diameter of the thoracic aorta (IVC / Ao) depends on the daily balance of fluids.

DETAILED DESCRIPTION:
During the routine abdominal ultrasound, the basilar and abdominal aorta were measured using a Sparq Philips ultrasonograph with a convex probe set in abdominal mode. All measurements were performed in one patient by the same operator who were experienced and performed the appropriate course of ultrasonography. The IVC and abdominal aorta were visualized using a paramedian long-axis view via a subcostal approach according to the methodology described by the American Society of Echocardiography. Inferior vena cava width was assessed at an interval of approximately 1 cm distal from connection of the hepatic vein to the inferior vena cava. No significant changes were observed in the width of the inferior vena cava during various respiratory phases, because of the positive pressure ventilation. The widest value was always chosen for the data. The assessment of the width of the abdominal aorta was performed above arise of the celiac trunk, at the height of the vein of the lower vena cava. The width of the inferior vena cava and the abdominal aorta was assessed using transthoracic ultrasound for the following five days. Daily differences in the amount of fluid intake and lost was recorded. CVP measurement was performed.

ELIGIBILITY:
Inclusion Criteria:

* patients who were hospitalized in the Intensive Care Unit
* severe respiratory failure requiring mechanical ventilation

Exclusion Criteria:

* spontaneous breathing,
* severe vascular disease,
* increased intra-abdominal pressure,
* cardiac pacemaker
* cardioverter defibrillator

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There were 57 mechanically ventilated patients examined. 8 patients were excluded from the study because of spontaneous ventilation within 5 days of data collection. Two patients died during the study. Five patients failed to obtain satisfactory results of imaging of vascular structures during subsequent examination. Data from 42 patients were analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
fluid balance | 1 day
  the width of the vena cava and abdominal aorta was measured every day morning. The difference in in taken and excreted fluids

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Skladzien, Ph.D., Principal Investigator — Jagiellonian University
Locations (1):
- University Hospital, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
The assessment of the width of the abdominal aorta was performed above arise of the celiac trunk, at the height of the vein of the lower vena cava. The width of the inferior vena cava and the abdominal aorta was assessed using transthoracic ultrasound for the following five days. Daily differences in the amount of fluid intake and lost was recorded. CVP measurement was performed.